CLINICAL TRIAL: NCT00154713
Title: A Phase I/II Clinical Study of Immunotherapy for Advanced Colorectal Cancers Using CEA-Pulsed Dendritic Cells Mixed With Tetanus Toxoid and Subsequent IL-2 Treatment
Brief Title: Immunotherapy for Colorectal Cancers Using CEA-Pulsed Dendritic Cells and Subsequent IL-2 Treatment
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27MD02
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; dendritic cell; CEA; IL-2
MeSH Terms: conditions — Colorectal Neoplasms

INTERVENTIONS:
Biological: CEA pulsed dendritic cells

SUMMARY:
The specific aims of this study are as follows:

1. Primary endpoint: to evaluate the clinical responses of vaccinated patients.
2. Secondary endpoint: to evaluate the safety of this treatment and the immune responses against CEA before and after the treatment

DETAILED DESCRIPTION:
In this trial, we will immunize metastatic colorectal cancer patients with recombinant CEA-pulsed DCs mixed with tetanus toxoid by subcutaneous injection. Low dose IL-2 will be given subcutaneously following DC vaccination to boost the growth of T cells. We will adapt "Simon's optimal two-stage design" for this study. In the first stage, we will treat 12 patients to evaluate the safety of this new protocol. If there are no severe toxicities/side effects and there is at least one patient that had stable disease or better clinical response, then we will proceed to the second stage and treat additional 25 patients. We will follow the clinical outcome of these 37 patients. The immune responses against CEA before and after vaccination will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic colorectal cancer.
* Patients must have at least one measurable lesion.
* Patients'serum level of CEA must be higher than 5 times of the normal value
* Patients'disease must have failed chemotherapy with 5FU, CPT-11 or oxaliplatin.
* Patients who are unsuitable or refuse chemotherapy will be considered eligible for this trial.
* Patients'age must be 20 or greater.
* Patients'estimated life expectancy is more than 3 months.
* Patients must have adequate bone marrow function, defined as WBC >= 3500/mm3, neutrophil >= 1500/mm3, lymphocyte >= 1,000/mm3, and platelet >= 100,000/mm3.
* Patients must have adequate liver and renal function, defined as serum alanine transaminase (ALT) and aspartate transaminase (AST) =< 5 times normal, bilirubin =< 1.5 times normal range, and creatinine =< 2 times upper normal limit.
* All patients should have documentation of negative result of penicillin test.
* Women or men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent.

Exclusion Criteria:

* Patients who have central nervous system metastasis except for those whose CNS disease has been treated with radiotherapy and/or surgery and has been stable for at least two weeks
* Patients who have active acute or chronic infection (at the discretion of the investigator).
* Pregnant or breast-nursing women
* Patients who have active cardiac disease requiring therapy for failure, angina, arrythmia, or infarction within the preceding 6 months (exception: any patient whose cardiac failure is compensated on medications)
* Patients who have asthma
* Patients who have autoimmune disease such as inflammatory bowel disease, lupus erythematosus, ankylosing spondylitis, scleroderma, and multiple sclerosis
* Patients who have serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator)
* Patients who have other prior or concurrent malignancy except for in-situ-carcinoma of cervix or adequately treated basal cell carcinoma of skin.
* Patients who received chemotherapy, steroid or biologic treatment within 4 weeks prior to enrollment

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37
Dates: Start 2005-07; Study Completion 2005-07

PRIMARY OUTCOMES:
evaluate the clinical responses of vaccinated patients 6 weeks after the first injection

SECONDARY OUTCOMES:
evaluate the safety of this treatment and the immune responses against CEA before and after the treatment 6 weeks after the first injection

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Whang-Peng, M.D., Principal Investigator — National Health Research Institutes, Taiwan; Hui-Ju Ch'ang, M.D., Principal Investigator — National Health Research Institutes, Taiwan; Ann-Li Cheng, M.D., Principal Investigator — National Taiwan University Hospital; Ko-Jiunn Liu, Ph.D., Principal Investigator — National Health Research Institutes, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Liu KJ, Chao TY, Chang JY, Cheng AL, Ch'ang HJ, Kao WY, Wu YC, Yu WL, Chung TR, Whang-Peng J. A phase I clinical study of immunotherapy for advanced colorectal cancers using carcinoembryonic antigen-pulsed dendritic cells mixed with tetanus toxoid and subsequent IL-2 treatment. J Biomed Sci. 2016 Aug 24;23(1):64. doi: 10.1186/s12929-016-0279-7. PMID 27558635